CLINICAL TRIAL: NCT06824376
Title: Efficacy and Safety Study of Manual Acupuncture (MA) on Serum Uric Acid (SUA) Outcomes in Patients With Asymptomatic Hyperuricemia (HUA): a Multi-center, Randomized, Sham-controlled Trial
Brief Title: Manual Acupuncture (MA) for Asymptomatic Hyperuricemia (HUA)
Acronym: HUA，SUA，MA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenghao Tu (Other)
Collaborators: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Xianning Hospital of Traditional Chinese Medicine, China (Unknown); Beijing Hospital of Traditional Chinese Medicine (Other); Qianjiang Central Hospital, China (Unknown); Hainan General Hospital (Other); Yichang Central People's Hospital (Other); Wuhan No.1 Hospital (Other); The Second Hospital of Huangshi (Unknown); Puyang Hospital of Traditional Chinese Medicine (Unknown)
Responsible Party: Sponsor-Investigator, Shenghao Tu, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023HUATJ01-V1.1(20240206); ZY2021Z002 (Other Grant/Funding Number: TCM Scientific Research Project of Hubei Provincial Health Commission)
Record Dates: First submitted 2025-01-14; First posted 2025-02-13 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Asymptomatic Hyperuricemia
Keywords: MA; HUA; SUA; deqi

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Manual acupuncture group (Experimental): Acupuncturists will apply 20 sessions of 30-mintute manual acupuncture at 10 obligatory acupoints, over 8 weeks of treatment period.
  Interventions: Device: Manual acupuncture
- Sham acupuncture group (Sham Comparator): 20 sessions of non-penetrating sham acupuncture will be performed at non-acupuncture points, which are located on the back and with different segments from the kidney organ area，over 8 weeks of treatment period.
  Interventions: Device: Sham acupuncture

INTERVENTIONS:
Device: Manual acupuncture — After sterilisation, the sharp needles will be inserted into the deep tissue layers of acupoints. Acupuncturists will tried to elicit acupuncture de-qi sensation by the manual manipulation of needles. Within a 30-minute period, manual manipulation for each acupoint will last at least 10 seconds and wil repeated four times with intervals of 10-minute.
  Arms: Manual acupuncture group
Device: Sham acupuncture — After sterilisation, Streitberger placebo needles with blunt tip will be used. It can be fixed on the surface of the sham points without piercing the skin. Within a 30-minute period, each point will undergo a simulated twisting motion of the needle for at least 10 seconds, and this will be repeated four times at 10-minute intervals.
  Arms: Sham acupuncture group

SUMMARY:
Assess the effectiveness of manual acupuncture in modulating serum uric acid levels among patients diagnosed with asymptomatic hyperuricemia.

DETAILED DESCRIPTION:
This is a multicenter randomized, single-blind, sham-controlled trial. A total of 260 eligible patients with asymptomatic hyperuricemia will be randomly assigned in a 1:1 ratio to manual acupuncture group or sham acupuncture group.

ELIGIBILITY:
Inclusion Criteria:

* With serum uric acid (SUA) level >7 mg/dL after 1 month of a low-purine diet.
* No history of gouty arthritis.
* Has not received uric acid-lowering drug treatment or stopped uric acid- lowering drug treatment ≥ 12 weeks.
* 18.5kg/m2 ≤ body mass index (BMI) ≤ 30.0 kg/m2.
* Can write informed consent.

Exclusion Criteria:

* Patients with poorly controlled hypertension: systolic blood pressure (SBP) ≥ 160mmHg, diastolic blood pressure (DBP) ≥ 100 mmHg.
* Patients with poorly controlled diabetes (hemoglobin A1c ≥ 8.4%).
* Patients with severe liver and kidney damage: chronic kidney disease (CKD) ≥ stage 2 or a serum creatinine, urea, alanine, or aspartate aminotransferase level more than twice of the upper limit.
* Patients with blood system diseases, such as acute and chronic leukemia, polycythemia, multiple myeloma, hemolytic anemia, lymphoma, or undergoing chemotherapy for multiple solid tumors.
* Patients with stroke, coronary heart disease, or severe neuropsychological diseases.
* Patients who are pregnant.
* Illiterate or unwilling to accept acupuncture treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Serum uric acid (SUA) | Baseline and 8 weeks after randomization.
  Changes in the SUA level after 8 weeks of treatment.

SECONDARY OUTCOMES:
Proportion of participants with SUA ≤ 6.0 mg/dL | 4 weeks after randomization, 8 weeks after randomization, 12 weeks after randomization and 16 weeks after randomization.
  The proportion of participants with SUA ≤ 6.0 mg/dL after treatment.
Proportion of participants with SUA ≤ 7.0 mg/dL. | 4 weeks after randomization, 8 weeks after randomization, 12 weeks after randomization and 16 weeks after randomization.
  The proportion of participants with SUA ≤ 7.0 mg/dL after treatment.
Dynamic changes in the SUA level after treatment. | Baseline, 4 weeks after randomization, 12 weeks after randomization and 16 weeks after randomization.
The proportion of participants with gout attacks | 4 weeks after randomization, 8 weeks after randomization, 12 weeks after randomization and 16 weeks after randomization.
  The proportion of participants with gout attacks after randomization

OTHER OUTCOMES:
Body weight | baseline, 4 weeks after randomization, 8 weeks after randomization, 12 weeks after randomization and 16 weeks after randomization.
  Changes in the body weight after treatment.
Abdominal circumference | baseline, 4 weeks after randomization, 8 weeks after randomization, 12 weeks after randomization and 16 weeks after randomization.
  Changes in abdominal circumference after treatment.
NEO Personality Inventory-Short Form (NEO-FFI) | baseline, 4 weeks after randomization, 8 weeks after randomization, 12 weeks after randomization and 16 weeks after randomization.
  NEO Personality Inventory-Short Form (NEO-FFI)
Traditional Chinese medicine (TCM) constitution | baseline, 4 weeks after randomization, 8 weeks after randomization, 12 weeks after randomization and 16 weeks after randomization.
  Changes in the Traditional Chinese medicine (TCM) constitution after treatment
Pittsburgh Sleep Quality Index (PSQI) | baseline, 4 weeks after randomization, 8 weeks after randomization, 12 weeks after randomization and 16 weeks after randomization.
  Changes in the PSQI after 4 weeks of treatment.
Beck Depression Inventory II (BDI- II) | baseline, 4 weeks after randomization, 8 weeks after randomization, 12 weeks after randomization and 16 weeks after randomization.
  Changes in the BDI- II after treatment.
Beck Anxiety Inventory (BAI) | baseline, 4 weeks after randomization, 8 weeks after randomization, 12 weeks after randomization and 16 weeks after randomization.
  Changes in the BAI after treatment
Adverse events (AEs) | From the beginning of acupuncture , up to 24 hours after acupuncture.
  AEs in which a causal relationship to the manual acupuncture or sham acupuncture cannot be ruled out will be considered an adverse reactions from the acupuncture. AEs related to acupuncture may include abnormal pain, bleeding, congestion, broken needles, bent needles, and dizziness.
The intensity of acupuncture de qi sensation. | Ten minutes after each manual or sham acupuncture treatment.
  The Massachusetts General Hospital (MGH) Acupuncture Sensation Scale (MASS) after each manual or sham acupuncture treatment

CONTACTS AND LOCATIONS:
Overall Officials: Shenghao Tu, Ph.D, Principal Investigator — Tongji Hospital
Locations (1):
- Institute of Integrated Traditional Chinese and Western Medicine, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
IPD after de-identification can be shared on individual request to the principal investigator at shtu@tjh.tjmu.edu.cn
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD and supporting information will be available after the publication of the primary outcomes.